CLINICAL TRIAL: NCT04655768
Title: Prospective Randomized Comparison of Conservative and Opertaive Treatment of Radius Fractures in Elderly Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kepler University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KUK-UNF-20-001
Record Dates: First submitted 2020-11-30; First posted 2020-12-07 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Orthopedic Disorder
Keywords: radius fracture, clinical outcome
MeSH Terms: conditions — Musculoskeletal Diseases; Radius Fractures

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Operative Arm (Active Comparator): Radius fractures C1/C2 treated by palmar plate fixation
  Interventions: Device: Palmar Plate Fixation
- Conservative Arm (No Intervention): Radius Fractures C1/C2 treated by cast fixation

INTERVENTIONS:
Device: Palmar Plate Fixation — Patients are treated by surgery (palmar plate)
  Arms: Operative Arm

SUMMARY:
Elderly Patients often suffer from radius fracture. Treatment options are conservative and operative. Aim of the stdy is to find out if there are diffrences in Patient's satisfaction depending on the different treatment.

A randomized prospective trial is palnned

DETAILED DESCRIPTION:
Patients of 70 years and more of age who suffer from C1 or C2 radius fracture are randomized treated by conservative treatment and operative treatment.

Primary aim is PRWE, secondary ROM as well as power and DASH score.

ELIGIBILITY:
Inclusion Criteria:

* Radius Fractures C1-C2
* age over 70

Exclusion Criteria:

* demetia
* collateral damages
* age < 70

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient Related Wrist Evaulation | 12-24 months post intervention
  PRWE, ROM investigation

SECONDARY OUTCOMES:
ROM | 12-24 months post intervention
  PRWE, ROM, Investigation

CONTACTS AND LOCATIONS:
Overall Officials: Stefan M Froschauer, MD, Study Director — Kepler University Hospital Linz
Locations (1):
- Kepler University Hospital, Linz, Upper Austria, Austria

IPD SHARING:
Plan to Share IPD: No